CLINICAL TRIAL: NCT02273154
Title: Randomized，Controlled and Open-label Study of Buspirone add-on Treatment in Patients With Major Depression Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Si Tianmei (Other)
Responsible Party: Sponsor-Investigator, Si Tianmei, Professor, Peking University
Organization: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUS-IV-01
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Major Depression Disorder
Keywords: major depressive disorder; Efficacy and safety of buspirone add-one treatment in patients with major depression disorder; buspirone; paroxetine; anxiety
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders | interventions — Buspirone; Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- paroxetine and buspirone group (Experimental): receive paroxetine (20-60mg/d) and buspirone(30mg/d)
  Interventions: Drug: Buspirone; Drug: Paroxetine
- paroxetine group (Active Comparator): receive paroxetine (20-60mg/d)
  Interventions: Drug: Paroxetine

INTERVENTIONS:
Drug: Buspirone — MDD patients with anxiety disorder take paroxetine (20-60mg/d), combining with buspirone (initial dose is 5mg tid, then increase the dose to 10mg tid on 4th day)
  Arms: paroxetine and buspirone group
Drug: Paroxetine — MDD patients with anxiety disorder take paroxetine (20-60mg/d)

SUMMARY:
This is a Multicenter, open lable, parallel randomized controlled clinical trial.

This study aimed to evaluate the treatment onset time, efficacy and safety in patients with major depressive disorders , accompanying anxiety receiving Buspirone and Paroxetine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meeting Statistical Manual of Mental Disorders IV (DSM-IV) criteria for major depression disorder , Hamilton Depression Rating Scale(HAM-D) score was 17 or above, Hamilton Anxiety Scale（HAMA）score was 7 or above.
2. aged 18-65 years( including 18,65 years )
3. male and female and inpatient as well as outpatient.
4. Written informed consent was obtained from each patient before therapy. -

Exclusion Criteria:

1. Patients with pregnant or breast-feeding and not taking effective contraceptive measures
2. Patients were allergic to buspirone or with a known intolerance to contraindication
3. Patients with clinically severe and unstable disease ,and not suitable to participate the study judged by the investigators
4. Patients with nervous system diseases(such as epilepsy, Brain injury, Multiple Sclerosis, Degenerative disease including acute lateral sclerosis, Parkinson's disease, ataxy)
5. Patients with a mental illness according to the DSM-IV, such as Organic mental disorders, Schizophrenia, Shizoaffective disorder, delusional disorder, Undifferentiated schizophrenia, bipolar disorder, and patients with a history of substance abuse including alcohol and active drug within 12 months of screening.
6. Patients are taking other Psychiatric drugs (such as Antipsychotic drugs, Anticonvulsant and Mood stabilizer but not include Antihistamine agents) and receiving ECT that might be excluded.
7. Patients worked on professional drivers or dangerous works
8. Patients participated in clinical trials within the past 30 days and treated with drugs from sponsors are not eligible.
9. Patients with clinically significant abnormalities on electrocardiogram or laboratory tests
10. Patients with Acute Angle-closure Glaucoma
11. Patients with Myasthenia Gravis
12. Patients who have used Monoamine oxidase inhibitors (MAOI) within 2 weeks of Screening
13. Patients who were Refractory depression invalid or non-responsive to adequate dosage (therapeutic dose upper limit) and duration (up 6 weeks) with two or above different antidepressants.
14. Patients who pose a suicidal risk, HAMD suicide score was 3 or above . -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Rate of onset of effect | 8 weeks
  defined as ≥20% change in HAMD total scores
clinical response rate | 8 weeks
  defined as ≥50% change in HAMD total scores
remission rate | 8 weeks
  Defined as HAMD total score ≤10.

SECONDARY OUTCOMES:
Changes of HAMD scores at week 4 and week 8 compared with baseline | 4 weeks
Changes of HAMA scores at week 4 and week 8 compared with baseline | 4 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Institute of mental health, Peking University, Beijing, Beijing Municipality
  - Henan mental health center, Xinxiang, Henan
  - Wuhan mental health center, Wuhan, Hubei
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - Dalian No.7 People's Hospital, Dalian, Liaoning
  - Shanxi Dayi Hospital, Taiyuan, Shanxi